CLINICAL TRIAL: NCT01353313
Title: A Randomized Controlled Trial of the Effect of Hydrocortisone on Survival Without Bronchopulmonary Dysplasia and on Neurodevelopmental Outcomes at 22 - 26 Months of Age in Intubated Infants < 30 Weeks Gestation Age
Brief Title: Hydrocortisone for BPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: National Center for Research Resources (NCRR) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NICHD-NRN-0045; U10HD034216 (NIH); U10HD027904 (NIH); U10HD021364 (NIH); U10HD027853 (NIH); U10HD040689 (NIH); U10HD040492 (NIH); U10HD027851 (NIH); U10HD021373 (NIH); U10HD027856 (NIH); U10HD053109 (NIH); U10HD036790 (NIH); U10HD027880 (NIH); U10HD053089 (NIH); U10HD021385 (NIH); U10HD068244 (NIH); U10HD068263 (NIH); U10HD068270 (NIH); U10HD068278 (NIH); U10HD068284 (NIH); U24HL137729 (NIH); 1UG3HL137872 (NIH)
Record Dates: First submitted 2011-04-20; First posted 2011-05-13 (Estimated); Results first posted 2022-08-19 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Infant, Newborn; Infant, Small for Gestational Age; Infant, Very Low Birth Weight; Infant, Premature; Bronchopulmonary Dysplasia
Keywords: NICHD Neonatal Research Network; Extremely Low Birth Weight (ELBW); Very Low Birth Weight (VLBW); Prematurity; Mechanical ventilation; Intubation; Neurodevelopmental impairment
MeSH Terms: conditions — Premature Birth; Bronchopulmonary Dysplasia | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Saline placebo
  Interventions: Drug: Placebo
- Hydrocortisone (Experimental): hydrocortisone sodium succinate for intravenous administration (unpreserved, Solu-Cortef plain, Pfizer®, reconstituted with unpreserved normal saline to avoid exposure to the benzyl alcohol contained in preserved diluents)
  Interventions: Drug: Hydrocortisone

INTERVENTIONS:
Drug: Hydrocortisone — Hydrocortisone sodium succinate for intravenous administration (unpreserved, Solu-Cortef plain, Pfizer®, reconstituted with unpreserved normal saline to avoid exposure to the benzyl alcohol contained in preserved diluents), to be administered either intravenously or orally if no intravenous line is available at the same dose, and tapered as follows:
  4mg/kg/day ¸ q 6 hours x 2 days, then 2mg/kg/day ¸ q 6 hours x 3 days; then
  1mg/kg/day ¸ q 12 hours x 3 days; then 0.5mg/kg/d as a single dose x 2 days
  Arms: Hydrocortisone
Drug: Placebo — Saline placebo to be administered either intravenously or orally if no intravenous line is available, at the same dose, and tapered as follows:
  4mg/kg/day ¸ q 6 hours x 2 days, then 2mg/kg/day ¸ q 6 hours x 3 days; then
  1mg/kg/day ¸ q 12 hours x 3 days; then 0.5mg/kg/d as a single dose x 2 days
  Arms: Placebo

SUMMARY:
The Hydrocortisone and Extubation study will test the safety and efficacy of a 10 day course of hydrocortisone for infants who are less than 30 weeks estimated gestational age and who are intubated at 14-28 days of life. Infants will be randomized to receive hydrocortisone or placebo. This study will determine if hydrocortisone improves infants'survival without moderate or severe BPD and will be associated with improvement in survival without moderate or severe neurodevelopmental impairment at 22 - 26 months corrected age.

DETAILED DESCRIPTION:
Bronchopulmonary dysplasia (BPD) remains a leading morbidity of the extremely preterm infant, and prolonged mechanical ventilation is associated with increased risk for BPD. Dexamethasone has been used previously to facilitate extubation and decrease the incidence of BPD; however, due to adverse effects on neurodevelopmental outcomes, the use of this drug has decreased. One cohort study suggests that hydrocortisone (HC) may facilitate extubation. HC has thus far not been associated with adverse neurodevelopmental outcomes in either cohort studies or randomized controlled trials. A recent meta-analysis of postnatal corticosteroid therapy begun after the first week of life suggested that "late therapy may reduce neonatal mortality without significantly increasing the risk of adverse long-term neurodevelopmental outcomes," although the methodological quality of some of the follow-up was acknowledged to be limited.

This is a randomized controlled trial to study the efficacy and safety of a 10-day tapering course of hydrocortisone treatment for infants <30 weeks estimated gestational age at birth who remain intubated at 14 - 28 days postnatal age. Based on previous Network data these criteria define a population with a risk of death or BPD at 36 weeks postmenstrual age of approximately 65 - 75%. The primary outcome for this study will incorporate both (1) survival without moderate to severe BPD by Network physiologic definition and (2) survival without moderate or severe NDI at 18 - 22 months corrected age. Therefore, the results of this study will be reported only when follow-up data are available unless (1) the trial is stopped early by the DSMC because of strong evidence of benefit or harm, or (2) at the time all subjects have completed treatment the DCC finds a substantial survival benefit favoring hydrocortisone (p<0.001). Individual study assignment will remain masked until the follow-up is completed. Secondary outcomes will include short term measures such as respiratory morbidities and growth at 36 weeks postmenstrual age and long term measures including growth and other outcomes at 22 - 26 months corrected age.

Secondary studies include:

1. Effect of Hydrocortisone on the Cardiac mass of Premature Intubated Infants - will determine left ventricular mass index at 36 weeks postmenstrual age (or prior to discharge/transfer if after 34 weeks) in infants enrolled in the hydrocortisone for BPD RCT, and compare HC-treated infants to placebo-treated infants. It will similarly assess and compare the incidence of pulmonary hypertension in these patients.
2. Extended follow-up: Subjects will be seen for a follow-up visit at 5-6 years corrected age to assess functional developmental and respiratory outcomes at early school age. In a subset of five Neonatal Research Network Clinical Centers, impulse oscillometry (IOS), which is the optimal direct measure of lung capacity and function, will be performed to validate the 6-minute walk test and International Study of Asthma and Allergies in Childhood (ISAAC) questionnaire as functional measures of pulmonary status. Also at these five Centers, the six minute walk test, ISAAAC questionnaire, and IOS will be administered as part of (1) the Healthy Lungs sub-study, which will recruit 120 TOP 5 study participants who had minimal lung disease when they were infants to define normative ranges in healthy, preterm-born children, and (2) the Healthy Lungs Two sub-study, which will recruit 120 healthy, term-born children without history of lung disease to characterize functional and mechanical respiratory outcomes at 5-7 years of age.

ELIGIBILITY:
Inclusion Criteria:

* infants <30 weeks estimated gestational age
* inborn at an NRN site or were admitted to an NRN site before 72 hours postnatal age
* have received at least 7days of mechanical ventilation;
* are receiving mechanical ventilation through an endotracheal tube .

Exclusion Criteria:

* Major congenital anomalies
* Decision to limit support
* Indomethacin or ibuprofen treatment within 48 hours of study drug
* Previous corticosteroid treatment for BPD
* Received hydrocortisone for 14 or more cumulative days
* Received hydrocortisone within 7 days of study entry

Max Age: 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 800 (Actual)
Dates: Start 2011-08-11 (Actual); Primary Completion 2020-09-21 (Actual); Study Completion 2024-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele C Walsh, MD, Principal Investigator — Case Western Reserve University, Rainbow Babies and Children's Hospital; Seetha Shankaran, MD, Principal Investigator — Wayne State University; Abbot R Laptook, MD, Principal Investigator — Brown University, Women & Infants Hospital of Rhode Island; C. Michael Cotten, MD, Principal Investigator — Duke University; David Carlton, MD, Principal Investigator — Emory University; Greg Sokol, MD, Principal Investigator — Indiana University; Abhik Das, PhD, Principal Investigator — RTI International; Krisa P Van Meurs, MD, Principal Investigator — Stanford University; Brenda P Poindexter, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Waldemar A Carlo, MD, Principal Investigator — University of Alabama at Birmingham; Edward F Bell, MD, Principal Investigator — University of Iowa; Kristi L Watterberg, MD, Study Chair — University of New Mexico; Myra Wyckoff, MD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas; Jon E Tyson, MD, MPH, Principal Investigator — The University of Texas Health Science Center, Houston; Eric Eichenwald, MD, Principal Investigator — University of Pennsylvania; Carl T D'Angio, MD, Principal Investigator — University of Rochester; Uday Devaskar, MD, Principal Investigator — University of California, Los Angeles; Pablo J Sanchez, MD, Principal Investigator — Research Institute at Nationwide Children's Hospital; William Truog, MD, Principal Investigator — Children's Mercy Hospital Kansas City; Bradley Yoder, MD, Principal Investigator — University of Utah
Locations (20):
- United States (20):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California - Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Wayne State University, Detroit, Michigan
  - Children's Mercy Hospital, Kansas City, Missouri
  - University of New Mexico, Albuquerque, New Mexico
  - University of Rochester, Rochester, New York
  - RTI International, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Research Institute at Nationwide Children's Hospital, Columbus, Ohio
  - Univeristy of Pennsylvania, Philadelphia, Pennsylvania
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
NIH has had a long-standing policy to share and make available to the public the results and accomplishments of the activities that it funds. The NRN plans to share de-identified data after final publication in an NIH supported data repository such as the NICHD Data and Specimen Hub (https://dash.nichd.nih.gov)

REFERENCES:
- [Derived] DeMauro SB, Kirpalani H, Hintz S, Watterberg KL, Watson V, Lowe J, Shankaran S, Chawla S, Vohr B, Msall ME, D'Angio CT, Yoder BA, Lai K, Winter S, Colaizy TT, Merhar SL, Ziolkowski K, Bann CM, Trotta M, Newman JE, Walsh MC, Higgins RD, Cahill TE, Duncan AF, Wilson-Costello DE, Peralta-Carcelen M, Arnold H, Mosquera RA, Heyne RJ, Fuller J, McGowan EC, Cavanaugh B, Harmon HM, Maitre NL, Neel ML, Van Meurs KP, Richards LA, Kilbride HW, Hines AC, Natarajan G, Trembath A, Benninger KL, Kesavan K, Malcolm WF, Zanger D, Reynolds AM, Carlson M, Das A; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Hydrocortisone in Preterm Infants and School-Age Functional Outcomes: Follow-Up of a Randomized Clinical Trial. JAMA Pediatr. 2025 Dec 8:e254801. doi: 10.1001/jamapediatrics.2025.4801. Online ahead of print. PMID 41359352
- [Derived] DeMauro SB, Kirpalani H, Ziolkowski K, Hintz S, Watterberg K, Lowe J, Shankaran S, Chawla S, Vohr B, Msall M, D'Angio C, Yoder BA, Lai K, Winter S, Colaizy T, Merhar S, Bann CM, Trotta M, Newman J, Natarajan A, Das A. The HYdrocortisone for Bronchopulmonary Dysplasia Respiratory and Developmental (HYBRiD) outcomes study: protocol for a longitudinal cohort study. BMC Pediatr. 2024 Nov 14;24(1):737. doi: 10.1186/s12887-024-05198-9. PMID 39543521
- [Derived] Gentle SJ, Rysavy MA, Li L, Laughon MM, Patel RM, Jensen EA, Hintz S, Ambalavanan N, Carlo WA, Watterberg K; National Institute of Child Health and Human Development Neonatal Research Network. Heterogeneity of Treatment Effects of Hydrocortisone by Risk of Bronchopulmonary Dysplasia or Death Among Extremely Preterm Infants in the National Institute of Child Health and Human Development Neonatal Research Network Trial: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2023 May 1;6(5):e2315315. doi: 10.1001/jamanetworkopen.2023.15315. PMID 37256621
- [Derived] Watterberg KL, Walsh MC, Li L, Chawla S, D'Angio CT, Goldberg RN, Hintz SR, Laughon MM, Yoder BA, Kennedy KA, McDavid GE, Backstrom-Lacy C, Das A, Crawford MM, Keszler M, Sokol GM, Poindexter BB, Ambalavanan N, Hibbs AM, Truog WE, Schmidt B, Wyckoff MH, Khan AM, Garg M, Chess PR, Reynolds AM, Moallem M, Bell EF, Meyer LR, Patel RM, Van Meurs KP, Cotten CM, McGowan EC, Hines AC, Merhar S, Peralta-Carcelen M, Wilson-Costello DE, Kilbride HW, DeMauro SB, Heyne RJ, Mosquera RA, Natarajan G, Purdy IB, Lowe JR, Maitre NL, Harmon HM, Hogden LA, Adams-Chapman I, Winter S, Malcolm WF, Higgins RD; Eunice Kennedy Shriver NICHD Neonatal Research Network. Hydrocortisone to Improve Survival without Bronchopulmonary Dysplasia. N Engl J Med. 2022 Mar 24;386(12):1121-1131. doi: 10.1056/NEJMoa2114897. PMID 35320643
- See also: NICHD Neonatal Research Network site — http://neonatal.rti.org/
- See also: NICHD Pregnancy & Perinatology Branch — https://www.nichd.nih.gov/about/org/der/branches/ppb/Pages/overview.aspx

RESULTS

PARTICIPANT FLOW:
Groups:
- Hydrocortisone: Hydrocortisone sodium succinate administered intravenously or orally if no intravenous line was available, tapered over 10 days.
- Placebo: Saline placebo administered intravenously or orally if no intravenous line was available.
Period: Overall Study
Arm/Group | Hydrocortisone | Placebo
Started | 398 | 402
Completed Assessment for Neurodevelopmental Impairment | 321 | 318
Died After Discharge | 8 | 6
Died Before Discharge | 35 | 40
Survived to Discharge | 363 | 362
Completed (Complete data for Neurodevelopmental Impairment or died) | 364 | 364
Not Completed | 34 | 38
Not completed — Lost to Follow-up | 22 | 23
Not completed — Incomplete Follow-up or No Study Data | 12 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydrocortisone | Placebo | Total
Number analyzed (Participants) | 398 | 402 | 800
Age, Continuous [Mean (Standard Deviation); unit: weeks] — Age refers to the infant and is measured as gestational age in weeks
  weeks | 24.9 (2) | 24.9 (2) | 24.9 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 212 | 167 | 379
  Male | 186 | 235 | 421
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race
  Participants
    Black | 139 | 168 | 307
    Missing | 10 | 11 | 21
    Other | 18 | 17 | 35
    White | 231 | 206 | 437
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity
  Participants
    Hispanic or Latino | 66 | 60 | 126
    Not Hispanic or Latino | 326 | 337 | 663
    Unknown or Not Reported | 6 | 5 | 11
Infant Body Weight [Mean (Standard Deviation); unit: grams] — Weight of the infant at birth, in grams
  grams | 710.3 (162.7) | 720.4 (171.8) | 715.4 (167.3)
Maternal Education [Count of Participants; unit: Participants] — Maternal education categories
  Participants
    College degree/more | 66 | 69 | 135
    High school degree | 101 | 108 | 209
    Less than High school degree | 68 | 59 | 127
    Partial college | 78 | 85 | 163
    Unknown | 85 | 81 | 166

OUTCOME MEASURES:

1. Primary Outcome: Survival Without Moderate/Severe Physiologic Bronchopulmonary Dysplasia (BPD)
Description: Survival without moderate or severe physiologic BPD at 36 weeks postmenstrual age. Moderate or severe physiologic BPD is defined as a requirement for supplemental oxygen and/or positive airway pressure to maintain oxygen saturation greater than 90 percent. A room air challenge was performed for infants estimated to be receiving less than 0.30 FiO2 by nasal cannula.
Time Frame: From day of randomization to 36 weeks post menstrual age
Population: The analysis population includes all randomized infants with available data at hospital discharge.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 398 | 402
Participants
  Moderate/severe BPD or death | 332 | 349
  Survival without moderate/severe physiologic bronchopulmonary dysplasia (BPD) | 66 | 53

2. Primary Outcome: Survival Without Moderate/Severe Neurodevelopmental Impairment (NDI)
Description: Survival without moderate or severe neurodevelopmental impairment (NDI) at 22-26 months corrected age. NDI is defined as defined as any of: Bayley Scales of Infant and Toddler Development-III (Bayley-III) cognitive composite score less than 85 (standardized mean 100, SD 15, range 55-145) or motor composite score less than 85 (standardized mean 100, range 45-155) (lower scores indicating greater impairment), Gross Motor Function Classification System (GMFCS) level greater than or equal to II (on a scale from level I to V; I=normal and progressively higher levels indicate greater impairment), severe vision impairment in both eyes (consistent with refraction from less than 20 to 200), or bilateral hearing impairment with or without amplification (by report).
Time Frame: From day of randomization to 22-26 months corrected age
Population: The analysis population includes all randomized infants with available data at the two-year followup.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 358 | 360
Participants
  Moderate/severe NDI or death | 226 | 226
  Survival without moderate/severe neurodevelopmental impairment (NDI) | 132 | 134

3. Secondary Outcome: Number of Participants With Successful Extubation
Description: Successful extubation during the intervention period, defined as remaining extubated for greater than or equal to 1 week, including greater than or equal to 3 days after the last dose of study medication. An extubation attempt was required after 72 hours of study drug and 24 hours after meeting the following: FiO2 less than 0.40 to maintain a saturation of greater than or equal to 88 percent, mean airway pressure less than 8 cm H2O, and hemodynamically stable in the opinion of the clinical team.
Time Frame: From day of randomization to day 14 post randomization
Population: The analysis population includes all randomized infants with available data at hospital discharge.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 398 | 402
Participants
  Successful extubation | 178 | 135
  Unsuccessful or no extubation | 220 | 267

4. Secondary Outcome: Total Deaths Before Discharge
Description: Infant died before discharge home.
Time Frame: From day of randomization to Neonatal Research Network NRN infant status i.e., the first occurring of: discharge home, death, transfer, or 120 days following birth
Population: The analysis population includes all randomized infants with available data at hospital discharge.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 398 | 402
Participants
  Death before discharge | 35 | 40
  Survival to discharge | 363 | 362

5. Secondary Outcome: Number of Participants With Bronchopulmonary Dysplasia (BPD) Grade at 36 Weeks Postmenstrual Age
Description: BPD grade at 36 weeks postmenstrual age. BPD grades are defined as: 1. No support/room air; 2. Nasal cannula (NC) O2 less than or equal to 2L; 3. NC O2 greater than 2L or CPAP/NIPPV; 4. Invasive PPV
Time Frame: At 36 weeks postmenstrual age
Population: The analysis population includes all randomized infants with available data at hospital discharge.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 375 | 367
Participants
  Invasive PPV | 63 | 51
  NC O2 greater than 2L or CPAP/NIPPV | 152 | 159
  Nasal cannula O2 less than or equal to 2L | 120 | 124
  No support, room air | 40 | 33

6. Secondary Outcome: Days of Mechanical Ventilation to 36 Weeks Postmenstrual Age (PMA)
Description: Number of days on mechanical ventilation (using high frequency ventilator or conventional ventilator)
Time Frame: From birth to 36 weeks postmenstrual age
Population: The analysis population includes all randomized infants with available data at hospital discharge.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 368 | 368
Days | 37 [27 to 54] | 40 [30 to 55]

7. Secondary Outcome: Duration of Oxygen Supplementation up to Status
Description: Number of days of oxygen supplementation from birth to discharge home
Time Frame: From birth to Neonatal Research Network NRN infant status i.e., the first occurring of: discharge home, death, transfer, or 120 days following birth
Population: The analysis population includes all randomized infants with available data who survived up to hospital discharge.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 362 | 362
Days | 104.5 [84 to 120] | 104 [83 to 120]

8. Secondary Outcome: Length of Hospital Stay in Days Among Survivors to Discharge
Description: Number of days infant stayed in hospitals, among those who survived to discharge
Time Frame: From birth up to one year
Population: The analysis population includes all randomized infants with available data at hospital discharge.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 362 | 362
Days | 127.5 [104 to 158] | 125.5 [106 to 155]

9. Secondary Outcome: Number of Participants With Dexamethasone Given Before 36 Weeks Postmenstrual Age (PMA)
Description: Infant received dexamethasone anytime before 36 weeks postmenstrual age.
Time Frame: From birth to 36 weeks postmenstrual age
Population: The analysis population includes all randomized infants with available data at hospital discharge.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 379 | 377
Participants
  Dexamethasone given before 36 weeks PMA | 150 | 157
  Dexamethasone not given before 36 weeks PMA | 229 | 220

10. Secondary Outcome: Number of Participants With Normal/Mild, Moderate or Severe/Profound NDI
Description: Severity of neurodevelopmental impairment, defined as one or more of: Bayley Scales of Infant Development-III (Bayley-III) cognitive score <85 (standardized mean 100, SD 15, range 55-145), Bayley-III motor score <85 (standardized mean 100, range 45-155), Gross Motor Function Classification System (GMFCS) level ≥2, severe vision impairment in both eyes (consistent with refraction <20-200), or bilateral hearing impairment with or without amplification (by report).
  Bayley-III = Bayley Scales of Infant Development III (Cognitive score standardized mean 100, SD 15, range 55-145 motor score standardized mean 100, range 45-155; higher score indicates better performance (20))
Time Frame: At 22-26 months corrected age
Population: The analysis population includes all randomized infants with available data who survived up to the two-year followup.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 315 | 314
Participants
  Moderate | 98 | 98
  Normal/mild | 132 | 134
  Severe/profound | 85 | 82

11. Secondary Outcome: Number of Participants With Gross Motor Function Greater Than or Equal to Level 2
Description: Number of infants with Gross Motor Function Classification System (GMFCS) level greater than or equal to II (on a scale from level I to V; I=normal and progressively higher levels indicate greater impairment)
Time Frame: At 22-26 months corrected age
Population: The analysis population includes all randomized infants with available data who survived up to the two-year followup.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 331 | 329
Participants
  Gross motor function less than II | 283 | 288
  Gross motor function level II or greater | 48 | 41

12. Secondary Outcome: Number of Participants With Moderate-severe Cerebral Palsy
Description: Number of infants with moderate or severe grade of cerebral palsy. Cerebral Palsy was diagnosed when there were definite abnormalities observed in the neuromotor exam, and functional challenges as classified by GMFCS level, and classified as moderate if GMFCS level was II or III and severe if level IV or V (40).
Time Frame: At 22-26 months corrected age
Population: The analysis population includes all randomized infants with available data who survived up to the two-year followup.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 330 | 330
Participants
  Moderate or severe cerebral palsy | 41 | 33
  Not moderate or severe cerebral palsy | 289 | 297

13. Secondary Outcome: Number of Participants With Severe Hearing Impairment (by Report)
Description: Number of infants with bilateral hearing impairment with or without amplification (by report)
Time Frame: At 22-26 months corrected age
Population: The analysis population includes all randomized infants with available data who survived up to the two-year followup.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 328 | 327
Participants
  Not severe hearing impairment | 319 | 313
  Severe hearing impairment | 9 | 14

14. Secondary Outcome: Number of Participants With no/Some Functional Vision
Description: Number of infants with severe vision impairment in both eyes (consistent with refraction less than 20-200)
Time Frame: At 22-26 months corrected age
Population: The analysis population includes all randomized infants with available data who survived up to the two-year followup.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 330 | 330
Participants
  Not severe vision impairment | 325 | 321
  Severe vision impairment | 5 | 9

15. Secondary Outcome: Weight Growth Measure Following Extremely Preterm Birth
Description: This is measured as the weight Z-score at 36 weeks postmenstrual age. The Z-score is derived using Fenton growth curves, and follows a standardized normal distribution with a mean 0. A z-score of 0 designates average weight, and negative scores denote less than average weight.
Time Frame: At 36 weeks post-menstrual age
Population: The analysis population includes all randomized infants with available data between 35 and 37 weeks at discharge.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 366 | 363
Z-score | -1.68 (1.01) | -1.65 (0.98)

16. Secondary Outcome: Follow-up Weight Growth Measure Following Extremely Preterm Birth
Description: This is measured as the weight Z-score at 22-26 months corrected age. The Z-score is determined using the WHO weight-for-age chart, and is derived from a standardized normal distribution, where 0 designates average weight-for-age, and negative scores denote less than average weight-for-age.
Time Frame: At 22-26 months corrected age
Population: The analysis population includes all randomized infants with available data between 18 and 30 months at follow-up.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 319 | 316
Z-score | -0.51 (1.04) | -0.44 (1.15)

17. Secondary Outcome: Length Growth Measure Following Extremely Preterm Birth
Description: This is measured as the length Z-score at 36 weeks postmenstrual age. The Z-score is derived using Fenton growth curves, and follows a standardized normal distribution with a mean 0. A z-score of 0 designates average length, and negative scores denote less than average length.
Time Frame: At 36 weeks post-menstrual age
Population: The analysis population includes all randomized infants with available data between 35 and 37 weeks at discharge.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 340 | 340
Z-score | -2.33 (1.16) | -2.21 (1.14)

18. Secondary Outcome: Follow-up Length Growth Measure Following Extremely Preterm Birth
Description: This is measured as the length Z-score at 22-26 months corrected age. The Z-score is determined using the WHO length-for-age chart, and is derived from a standardized normal distribution, where 0 designates average length-for-age, and negative scores denote less than average length-for-age.
Time Frame: At 22-26 months corrected age
Population: The analysis population includes all randomized infants with available data between 18 and 30 months at follow-up.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 316 | 314
Z-score | -0.93 (1.17) | -0.94 (1.22)

19. Secondary Outcome: Head Circumference Growth Measure Following Extremely Preterm Birth
Description: This is measured as the head circumference Z-score at 36 weeks postmenstrual age. The Z-score is derived using Fenton growth curves, and follows a standardized normal distribution with a mean 0. A z-score of 0 designates average head circumference, and negative scores denote less than average head circumference.
Time Frame: At 36 weeks post-menstrual age
Population: The analysis population includes all randomized infants with available data between 35 and 37 weeks at discharge.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 353 | 354
Z-score | -1.68 (1.34) | -1.74 (1.17)

20. Secondary Outcome: Follow-up Head Circumference Growth Measure Following Extremely Preterm Birth
Description: This is measured as the head circumference Z-score at 22-26 months corrected age. The Z-score is determined using the WHO head circumference-for-age chart, and is derived from a standardized normal distribution, where 0 designates average head circumference-for-age, and negative scores denote less than average head circumference-for-age.
Time Frame: At 22-26 months corrected age
Population: The analysis population includes all randomized infants with available data between 18 and 30 months at follow-up.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 314 | 301
Z-score | -0.45 (1.41) | -0.35 (1.42)

21. Secondary Outcome: Number of Participants With Bronchopulmonary Dysplasia (BPD) Grade 40 Weeks Postmenstrual Age
Description: BPD grade at 40 weeks postmenstrual age. BPD grades are defined as: 1. No support/room air; 2. Nasal cannula (NC) O2 less than or equal to 2L; 3. NC O2 greater than 2L or CPAP/NIPPV; 4. Invasive PPV
Time Frame: At 40 weeks post menstrual age
Population: The analysis population includes all randomized infants with available data at hospital discharge.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 279 | 284
Participants
  Invasive PPV | 46 | 38
  NC O2 greater than 2L or CPAP/NIPPV | 73 | 65
  Nasal cannula O2 less than or equal to 2L | 124 | 129
  No support, room air | 36 | 52

22. Secondary Outcome: Days of Mechanical Ventilation up to Status
Description: Number of days on mechanical ventilation (using high frequency ventilator or conventional ventilator) up to status
Time Frame: as for outcome 7
Population: The analysis population includes all randomized infants with available data who survived up to hospital discharge.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 361 | 362
Days | 37 [27 to 56] | 41 [30 to 56]

23. Secondary Outcome: Duration of Oxygen Supplementation Among Survivors to 36 Weeks
Description: Number of days of oxygen supplementation from birth to 36 weeks post menstrual age
Time Frame: From birth to 36 weeks postmenstrual age
Population: The analysis population includes all randomized infants with available data at hospital discharge.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 369 | 368
Days | 74 [65 to 81] | 73 [64 to 82]

24. Secondary Outcome: Duration of Invasive Positive Pressure Ventilation (PPV) After Postnatal Day 14
Description: Number of days on invasive PPV after postnatal day 14
Time Frame: From postnatal day 15 to 36 weeks post menstrual age or Neonatal Research Network NRN infant status i.e., the first occurring of: discharge home, death, transfer, or 120 days following birth
Population: The analysis population includes all randomized infants with available data who were extubated prior to hospital discharge.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 161 | 124
Days | 29 [16 to 40] | 27 [16 to 34.5]

25. Secondary Outcome: Duration of Non-invasive Positive Pressure Ventilation (PPV) (Nasal IPPV/CPAP) After Postnatal Day 14
Description: Number of days of non-invasive PPV after postnatal day 14
Time Frame: as for outcome 24
Population: as for outcome 24
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 161 | 124
Days | 13 [8 to 18] | 13 [7 to 19]

26. Secondary Outcome: Number of Participants Who Received Inhaled Glucocorticoids During Study Period
Description: Number of infants who received Inhaled glucocorticoids during the study intervention period
Time Frame: From randomization to day 14 post randomization
Population: The analysis population includes all randomized infants with available data at hospital discharge.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 396 | 399
Participants
  Did not receive inhaled glucocorticoids during study period | 345 | 355
  Received inhaled glucocorticoids during study period | 51 | 44

27. Secondary Outcome: Number of Participants Who Received Other Systemic Glucocorticoids During Study Period
Description: Number of infants who received other systemic glucocorticoids during the study intervention period
Time Frame: From randomization to day 14 post randomization
Population: The analysis population includes all randomized infants with available data at hospital discharge.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 396 | 399
Participants
  Did not receive other systemic glucocorticoids during study period | 342 | 334
  Received other systemic glucocorticoids during study period | 54 | 65

28. Secondary Outcome: Number of Days Dexamethasone Given Before 36 Weeks PMA
Description: Number of days infant received dexamethasone anytime before 36 weeks postmenstrual age.
Time Frame: From birth to 36 weeks postmenstrual age
Population: The analysis population includes all randomized infants with available data at hospital discharge.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 150 | 157
Days | 10 [8 to 12] | 10 [4 to 11]

29. Secondary Outcome: Number of Participants With Patent Ductus Arteriosus (PDA) Treated With Medication or Surgery
Description: Number of infants with a Patent Ductus Arteriosus (PDA) that was treated with medicine or surgery
Time Frame: as for outcome 7
Population: The analysis population includes all randomized infants with available data at hospital discharge.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 398 | 402
Participants
  Not PDA treated with medication or surgery | 206 | 209
  PDA treated with medication or surgery | 192 | 193

30. Secondary Outcome: Number of Participants Diagnosed With Necrotizing Enterocolitis (NEC)
Description: Number of infants diagnosed with Necrotizing Enterocolitis (NEC)
Time Frame: as for outcome 7
Population: The analysis population includes all randomized infants with available data at hospital discharge.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 398 | 402
Participants
  Diagnosed with NEC | 33 | 46
  Not diagnosed with NEC | 365 | 356

31. Secondary Outcome: Number of Participants With Retinopathy of Prematurity (ROP) Stage 3 or Worse
Description: Number of infants diagnosed with ROP stage 3 or worse in either eye. ROP stage 3 or worse is determined based on the extent of extraretinal fibrovascular proliferation. Higher stages of ROP indicate a worse outcome; the stages range from 1 for "mild" disease, to 5 for "severe" disease.
Time Frame: as for outcome 7
Population: The analysis population includes all randomized infants with available data at hospital discharge.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 382 | 376
Participants
  Diagnosed with ROP stage 3 or worse | 105 | 116
  Not diagnosed with ROP stage 3 or worse | 277 | 260

32. Secondary Outcome: Number of Participants Receiving Therapy for Retinopathy of Prematurity (ROP)
Description: Number of infants receiving therapy for Retinopathy of prematurity (ROP)
Time Frame: as for outcome 7
Population: The analysis population includes all randomized infants with available data at hospital discharge.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 379 | 376
Participants
  Did not receive therapy for ROP | 311 | 293
  Received therapy for ROP | 68 | 83

33. Secondary Outcome: Number of Participants With Severe Intraventricular Hemorrhage (IVH)
Description: Number of infants with severe IVH, grade 3 or 4. Severity of IVH is hierarchical. Grade 3 occurs when the ventricular size is enlarged and blood/echodensity is in the ventricle. Grade 4 occurs when blood/echodensity is in the parenchyma.
Time Frame: as for outcome 7
Population: The analysis population includes all randomized infants with available data at hospital discharge.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 397 | 402
Participants
  Not severe IVH, grade 3 or 4 | 316 | 331
  Severe IVH, grade 3 or 4 | 81 | 71

34. Secondary Outcome: Number of Participants With Periventricular Leukomalacia
Description: Number of infants with Periventricular leukomalacia
Time Frame: as for outcome 7
Population: The analysis population includes all randomized infants with available data at hospital discharge.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 398 | 402
Participants
  No periventricular leukomalacia | 376 | 378
  Periventricular leukomalacia | 22 | 24

35. Secondary Outcome: Number of Participants With Neurodevelopmental Impairment (NDI)
Description: Number of infants with NDI. NDI is defined as defined as any of: Bayley Scales of Infant and Toddler Development-III (Bayley-III) cognitive composite score less than 85 (standardized mean 100, SD 15, range 55-145) or motor composite score less than 85 (standardized mean 100, range 45-155) (lower scores indicating greater impairment), Gross Motor Function Classification System (GMFCS) level greater than or equal to II (on a scale from level I to V; I=normal and progressively higher levels indicate greater impairment), severe vision impairment in both eyes (consistent with refraction less than 20-200), or bilateral hearing impairment with or without amplification (by report).
Time Frame: At 22-26 months corrected age
Population: The analysis population includes all randomized infants with available data at the two-year followup.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 321 | 319
Participants
  Neurodevelopmental impairment | 189 | 185
  No neurodevelopmental impairment | 132 | 134

36. Secondary Outcome: Number of Participants With a Bayley Scales of Infant Development (BSID) Cognitive Composite Score Less Than 85
Description: Number of infants with a BSID-III cognitive composite score less than 85. (standardized mean 100, SD 15, range 55-145). Higher scores indicate better performance. Composite BSID-III scores of less than 85 are less than 1 standard deviation below the mean of 100.
Time Frame: At 22-26 months corrected age
Population: The analysis population includes all randomized infants with available data at the two-year followup.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 318 | 318
Participants
  Composite cognitive score greater or equal to 85 | 168 | 176
  Composite cognitive score less than 85 | 150 | 142

37. Secondary Outcome: Number of Participants With a Bayley Scales of Infant Development (BSID) Cognitive Composite Score Less Than 70
Description: Number of infants with a BSID-III cognitive composite score less than 70. (standardized mean 100, SD 15, range 55-145). Composite BSID-III scores of less than 70 are less than 2 standard deviations below the mean of 100.
Time Frame: At 22-26 months corrected age
Population: The analysis population includes all randomized infants with available data at the two-year followup.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 318 | 318
Participants
  Composite cognitive score greater or equal to 70 | 259 | 269
  Composite cognitive score less than 70 | 59 | 49

38. Secondary Outcome: Number of Participants With a Bayley Scales of Infant Development (BSID) Motor Composite Score Less Than 85
Description: Number of infants with a BSID-III motor composite score less than 85. (standardized mean 100, SD 15, range 55-145). Composite BSID-III scores of less than 85 are less than 1 standard deviation below the mean of 100.
Time Frame: At 22-26 months corrected age
Population: The analysis population includes all randomized infants with available data at the two-year followup.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 310 | 310
Participants
  Composite motor score greater or equal to 85 | 164 | 158
  Composite motor score less than 85 | 146 | 152

39. Secondary Outcome: Number of Participants With a Bayley Scales of Infant Development (BSID) Motor Composite Score Less Than 70
Description: Number of infants with a BSID-III motor composite score less than 70. (standardized mean 100, SD 15, range 55-145). Composite BSID-III scores of less than 70 are less than 2 standard deviations below the mean of 100.
Time Frame: At 22-26 months corrected age
Population: The analysis population includes all randomized infants with available data at the two-year followup.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 310 | 310
Participants
  Composite motor score greater or equal to 70 | 241 | 246
  Composite motor score less than 70 | 69 | 64

40. Secondary Outcome: Number of Participants With Any Cerebral Palsy
Description: Number of infants with cerebral palsy. Cerebral Palsy was diagnosed when there were definite abnormalities observed in the neuromotor exam, and functional challenges as classified by GMFCS level, and classified as moderate if GMFCS level was II or III and severe if level IV or V (40).
Time Frame: At 22-26 months corrected age
Population: The analysis population includes all randomized infants with available data at the two-year followup.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 330 | 330
Participants
  Any cerebral palsy | 84 | 71
  No cerebral palsy | 246 | 259

ADVERSE EVENTS:
Time Frame: Birth to 36 weeks PMA
Arm/Group | Hydrocortisone | Placebo
All-Cause Mortality (participants affected / at risk) | 43/398 | 46/402
Serious Adverse Events (participants affected / at risk) | 84/398 | 95/402
Other Adverse Events (participants affected / at risk) | 106/398 | 95/402
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hydrocortisone (N=398) | Placebo (N=402)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Adrenal insufficiency neonatal (Congenital, familial and genetic disorders) | 5 | 16
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 1 | 4
Abdominal compartment syndrome (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 9 | 13
Lip ulceration (Gastrointestinal disorders) | 1 | 0
Necrotizing enterocolitis neonatal (Gastrointestinal disorders) | 2 | 5
Necrotizing enterocolitis neonatal (Totalis) (Gastrointestinal disorders) | 0 | 1
Liver injury (Hepatobiliary disorders) | 1 | 0
Nosocomial infection (Infections and infestations) | 32 | 29
Osteomyelitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 6 | 2
Pneumonia (MRSA) (Infections and infestations) | 1 | 0
Sepsis neonatal (Infections and infestations) | 2 | 3
Septic shock (Infections and infestations) | 1 | 1
Ureaplasma infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 1
Extra-axial hemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 28 | 19
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 4
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 2
Rickets (Musculoskeletal and connective tissue disorders) | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 1
Hydrops foetalis (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 2
Acute renal failure (Renal and urinary disorders) | 0 | 1
Anuria (Renal and urinary disorders) | 0 | 1
Oliguria (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 61 | 61
Hypertension (Vascular disorders) | 15 | 4
Hypotension (Vascular disorders) | 2 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 0.05% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Hydrocortisone (N=398) | Placebo (N=402)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 2
Tachycardia (Cardiac disorders) | 1 | 0
Adrenal insufficiency neonatal (Congenital, familial and genetic disorders) | 22 | 24
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 5 | 5
Necrotizing enterocolitis neonatal (Suspected) (Gastrointestinal disorders) | 0 | 1
Bacterial disease carrier (Infections and infestations) | 1 | 0
Nosocomial infection (Infections and infestations) | 18 | 27
Pneumonia (Infections and infestations) | 1 | 3
Pneumonia mycoplasmal (Infections and infestations) | 0 | 1
Sepsis neonatal (Infections and infestations) | 5 | 7
Tracheitis (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 0 | 3
Wound infection (Neck) (Infections and infestations) | 1 | 0
Alkaline phosphatase NOS increased (Investigations) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 25 | 12
Hyperkalemia (Metabolism and nutrition disorders) | 5 | 6
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 4 | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 1
Oliguria (Renal and urinary disorders) | 2 | 0
Prerenal failure (Renal and urinary disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 41 | 48
Hypertension (Vascular disorders) | 56 | 29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators must adhere to the Neonatal Research Network Publication Policies

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2013-08-27): https://cdn.clinicaltrials.gov/large-docs/13/NCT01353313/Prot_SAP_000.pdf
  • Informed Consent Form (2012-05-07): https://cdn.clinicaltrials.gov/large-docs/13/NCT01353313/ICF_001.pdf